CLINICAL TRIAL: NCT06499922
Title: Recent Advances in Surgical Management of Low Grade Glioma
Brief Title: Surgical Management of Low Grade Glioma
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, M.Hossam Mohammad, principal investigator, Assiut University
Other Study IDs: Surgery of low grade glioma
Record Dates: First submitted 2024-05-31; First posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Low Grade Glioma of Brain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: SURGICAL EXCISION — surgical excision of low grade glioma

SUMMARY:
To assess the morbidity and mortality in low grade glioma patients following surgical management.

DETAILED DESCRIPTION:
lower-grade gliomas histological diagnosis has had a long history, each iteration of disease classification suffered from continued variability, with detrimental consequences on prognostic precision and treatment decision making.

In the WHO 2021 classification, there are three primary categories of adult-type diffuse gliomas: isocitrate dehydrogenase (IDH)-mutant, 1p/19q codeleted oligodendroglioma; IDH-mutant, non-codeleted astrocytoma; and IDH-wildtype glioblastoma. Diffuse low-grade glioma is classified as WHO grade 1 and 2 astrocytoma with IDH mutation or oligodendroglioma with IDH mutation and 1p/19q codeletion.

The presence of the IDH1 mutation has become a defining factor for adult diffuse low-grade glioma. Roughly 70% of grade 2-3 gliomas harbor mutations in either IDH1 or its mitochondrial counterpart IDH2.

Although lower-grade gliomas may present in various ways, the most common manifestation is seizures, and the development of seizures during the course of the disease may herald tumor progression. Among grade II tumors, the incidence of epilepsy is higher with IDH mutation. Anaplastic gliomas are somewhat less likely to manifest with seizures (57%) and are more likely than grade II gliomas to produce mental status, vision, and motor deficits.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed radiologically with low grade glioma

Exclusion Criteria:

* patients not fit for surgery

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Each patient will be subjected to:
  * A complete history including personal history, history of seizures or drug intake.
  * General clinical examination.
  * Neurological examination.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Morbidity in low grade glioma patients following surgical management. | 2 years
  report THE RATE OF POSTOPERATIVE MORBIDITY Among participants using the neurological condition assessment ( kornofisky Scale).

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed El Gheriani, professor, Study Chair — professor

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Davis ME. Epidemiology and Overview of Gliomas. Semin Oncol Nurs. 2018 Dec;34(5):420-429. doi: 10.1016/j.soncn.2018.10.001. Epub 2018 Nov 2. PMID 30392758
- [Background] Louis DN, Perry A, Wesseling P, Brat DJ, Cree IA, Figarella-Branger D, Hawkins C, Ng HK, Pfister SM, Reifenberger G, Soffietti R, von Deimling A, Ellison DW. The 2021 WHO Classification of Tumors of the Central Nervous System: a summary. Neuro Oncol. 2021 Aug 2;23(8):1231-1251. doi: 10.1093/neuonc/noab106. PMID 34185076
- [Background] Mazzucchi E, La Rocca G, Ius T, Sabatino G, Della Pepa GM. Multimodality Imaging Techniques to Assist Surgery in Low-Grade Gliomas. World Neurosurg. 2020 Jan;133:423-425. doi: 10.1016/j.wneu.2019.10.120. No abstract available. PMID 31881559